CLINICAL TRIAL: NCT05627843
Title: Effects of Curcumin on Inflammation and Oxidative Stress in Paediatric Patients on Regular Hemodialysis: A Randomized, Double-Blind, Placebo-Controlled Pilot Study
Brief Title: Effects of Curcumin on Inflammation and Oxidative Stress in Pediatric Patients on Regular Hemodialysis: A Randomized, Double-Blind, Placebo-Controlled Pilot Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Mohamed Naguib Alagamy, Assistant lecturer at Misr university for science and technology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD 181 / 2021
Record Dates: First submitted 2022-11-02; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Pediatric Patients Having Renal Failure and on Regular Hemodialysis
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): Children on regular hemodialysis whose weight 30 kg or above
  Interventions: Dietary Supplement: Curcumin capsules 1 gm
- Placebo group (Placebo Comparator): Children on regular hemodialysis whose weight 30 kg or above
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Curcumin capsules 1 gm — Dietary supplement
  Arms: Trial group
Dietary Supplement: Placebo capsule — placebo corn starch
  Arms: Placebo group

SUMMARY:
* The study will be a randomised, double blinded, placebo controlled design.
* It will include 2 groups : trial group and placebo group
* Patients in both groups are children on regular hemodialysis
* The patients in the trial group will receive Curcumin capsule 1 gm for 3 months , and the placebo group will receive a placebo capsule for 3 months
* All patients will be evaluated clinically, and laboratory at baseline, at 3 months after end of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric patients with weight of at least 30 kilograms.
* Undergoing regular hemodialysis for at least 6 months.

Exclusion Criteria:

* Bleeding disorders.
* Chronic liver disease.
* Diabetes mellitus.
* Autoimmune diseases.
* Receiving drugs that are contraindicated, or have major interactions with curcumin, and can't be discontinued or replaced.
* Receiving corticosteroids, or immune-suppressants.
* Patients taking any antioxidant supplements including vitamin E, ascorbic acid, omega -3 fatty acid, or L-carnitine within 3 months prior to enrollment in our study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
inflammatory marker | 3 months
  high sensitivity C reactive protein (CRP) at baseline before supplementation and after 3 months of supplementation

SECONDARY OUTCOMES:
Oxidative stress markers | 3 months
  Serum tumor necrotizing factor alpha (TNF alpha)and malondialdehyde (MDA)at baseline and after 3 months of supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Iman Mohamed Naguib Alagamy, Cairo, Egypt